CLINICAL TRIAL: NCT07361939
Title: Evaluation of the Safety and Effectiveness of easyEndoTM Lite Linear Cutting Stapler and Loading Unit in Gastrointestinal Surgery: a Retrospective, Observational, Post Market Study
Brief Title: easyEndoTM Lite Stapler Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ezisurg Medical Co. Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lite-T
Record Dates: First submitted 2025-12-17; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- easyEndoTM Lite Linear Cutting Stapler and staggered design Loading Unit (Experimental)
  Interventions: Device: easyEndoTM Lite Linear Cutting Stapler and staggered design Loading Unit

INTERVENTIONS:
Device: easyEndoTM Lite Linear Cutting Stapler and staggered design Loading Unit — The Staplers are available in 260mm, 350mm and 440mm lengths. Loading Units for Single Use are available in eight staple sizes to accommodate various tissue thickness: 2.0mm, 2.5mm, 3.5mm, 3.8mm, 4.1mm, 2.0-2.5-3.5mm and 3.5-3.8-4.1mm, 3.8-4.1-4.4mm.

SUMMARY:
The purpose of this observational study is to evaluate the safety and performance of the easyEndoTM Lite Linear Cutting Stapler and staggered design Loading Unit from EziSurg Medical in gastrointestinal surgery. The goal of the study will be achieved by assessing the device performance and reporting of peri- and postoperative complications retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Age at study entry is at least 18 years.
* The operation involves the application of easyEndoTM Lite Stapler and Loading Unit for tissue cutting and suturing.

Exclusion Criteria:

* Pregnancy.
* Emergency operation (such as acute intestinal obstruction and gastrointestinal perforation).
* Assessed by the investigator, whose condition is poor and cannot tolerate the surgery.
* History of gastrointestinal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
stapling success rate | Perioperative/Periprocedura

SECONDARY OUTCOMES:
postoperative complications | Perioperative/Periprocedural
Technical success rate | Perioperative/Periprocedural
  defined as completion of gastrointestinal surgery as intended without technical difficulties and/or without conversion to open laparotomy

CONTACTS AND LOCATIONS:
Locations (1):
- Saida Center, Lebanon, Beirut, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: No